CLINICAL TRIAL: NCT05075551
Title: Analyzing the Brain Alterations of Acupuncture on Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome Evaluated by fMRI: Study Protocol for a Randomized Trial
Brief Title: Analyzing the Brain Alterations of Acupuncture on Patients With CP/CPPS Evaluated by fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 681328
Record Dates: First submitted 2021-09-19; First posted 2021-10-12 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Chronic Prostatitis/Chronic Pelvic Pain Syndrome; Functional Magnetic Resonance Imaging; Acupuncture
MeSH Terms: conditions — Prostatitis | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The eligible participants will receive either acupuncture or sham acupuncture randomly assigned at the ratio of 1:1 after signing the Informed consent. Before they accept the treatment, they are acquired to finish the clinical scales and get the fMRI scan. Sanyinjiao (SP6), Zhibian (BL54), Shenshu (BL23), and Huiyang (BL35) have been chosen as acupoints. In the group of both acupuncture and sham acupuncture, the course of treatment is 2 times a week in three months (totally 24 times). There are 3 clinic visits and 3 telephone contacts for emergency. At the ending of the treatment, all the volunteers will be asked to finish the clinical scales and get the fMRI scan again. As the step of following up, all the patients will be asked to finish the clinical scales and get the fMRI scan again to evaluate the efficacy of avoiding the recurrence of acupuncture.
Who Masked: Participant, Outcomes Assessor
Masking Description: Owing to differentiating the acupuncture effect from placebo effect, the participants and outcomes assessors are needed to be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Before participants accept the treatment, they are acquired to finish the clinical scales (including NIH-CPSI scale, HADS, VAS, SSRS, SES, IPSS and QoL) and then get the fMRI scan. Hwato brand disposable acupuncture needles will be used. Sanyinjiao (SP6), Zhibian (BL54), Shenshu (BL23), and Huiyang (BL35) are selected as acupoints. The course of treatment is 2 times a week in three months (totally 24 times). At the ending of the treatment, all the volunteers will be asked to finish the clinical scales and get the fMRI scan again. As the step of following up, all the patients will be asked to finish the clinical scales and get the fMRI scan again to evaluate the efficacy of avoiding the recurrence of acupuncture.
  Interventions: Device: Acupuncture; Other: fMRI scan
- Sham Acupuncture (Sham Comparator): In the sham acupuncture group, these volunteers will receive relatively shallow needling at bilateral sham SP6, BL54, BL23, and BL35. This treatment gets involved in the same duration and frequency of sessions, but the treatment was delivered superficially at non-acupuncture points 10 mm to the lateral of corresponding acupuncture and not above a meridian line (10mm to SP6, BL54, BL23 and BL35). The Hwato brand disposable acupuncture needles will be inserted with a depth of 2-3 mm without any manipulation.The procedure of finishing scales and get fMRI scanning will be the same as the group of acupuncture.
  Interventions: Device: Sham acupuncture; Other: fMRI scan

INTERVENTIONS:
Device: Acupuncture — Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used.SP6 is on the tibial aspect of the leg, posterior to the medial border of the tibia, 3 cun superior to the prominence of the medial malleolus; BL23 is in the sacral region, in the second posterior sacral foramen; BL54 is in the fourth posterior sacral foramen, 3 cun beside the median sacral crest; BL35 is in the buttock region, 0.5 cun lateral to the extremity of the coccyx.
  Arms: Acupuncture
Device: Sham acupuncture — Hwato brand disposable acupuncture needles (size 0.30 × 75mm; size 0.30 × 40mm) will be used.These volunteers will receive relatively shallow needling at bilateral sham SP6, BL54, BL23 and BL35. This treatment gets involved in the same duration and frequency of sessions, but the treatment was delivered superficially at non-acupuncture points 10 mm to the lateral of corresponding acupuncture and not above a meridian line (10mm to SP6, BL54, BL23 and BL35).The same equipment of fMRI scanner will be used.
  Arms: Sham Acupuncture
Other: fMRI scan — Both two group will get fMRI scan week 0 (before treatment), week 12 (after treatment) and week 36 (following up). The resting-state fMRI data will be obtained by using a 3.0T GE MR 750 MRI scanner with an eight-channel phase array head coil at the Huashan Hospital, Shanghai. The high resolution T1-weighted magnetic resonance images will be collected by a three-dimensional fast spoiled gradient-echo dual-echo sequence [repetition time (TR) = 8100 ms; echo time (TE) = 3.1 ms; FA = 8 deg; matrix=256 × 256; field of view (FOV)=25.6× 25.6 cm2; slice thickness=1 mm; no gap and 156 slices]. The whole resting state fMRI data will be acquired by using a gradient-recalled echo-planar imaging pulse sequence (TR/TE = 2,000/30 ms; FA = 90°; acquisition matrix = 64×64; FOV = 22×22 cm2; slice thickness= 4 mm; 43 slices and total 240 time points; no gap).

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is one of the most common diseases in urology, but its pathogenesis remains unclear and the effective therapy lacks. As a kind of chronic pain which the patients suffered for more than 3 months, CP/CPPS could be alleviated by acupuncture. Functional magnetic resonance imaging (fMRI) and higher magnetic field strengths could enable scientists to investigate the brain accurately and non-invasively during every stage of chronic pain.To avoid placebo effect, sham acupuncture would be also enrolled.Herein, by the utilization of fMRI in resting-state, we investigated the influence on patients' brain alterations after the patients accepted the treatment of acupuncture.

DETAILED DESCRIPTION:
A two (participant and assessor) blind, two-arm parallel, randomized controlled trial will be conducted. Sixty patients with CP/CPPS will be recruited from Huashan Hospital, Shanghai, and thirty healthy volunteers will be recruited as the healthy control group by advertisement. Patients will be randomly assigned into one of two intervention groups: acupuncture group and sham acupuncture group. The ratio of healthy control (n = 30), acupuncture group (n = 30) and sham acupuncture group (n = 30) will be 1:1:1. Sanyinjiao (SP6), Zhibian (BL54), Shenshu (BL23), and Huiyang (BL35) are chosen as acupoints for both acupuncture group and sham acupuncture group (Park sham device). The course of treatment is 2 times a week in three months (totally 24 times). The group of healthy control will get only once fMRI scan while the group of patients will get fMRI scan week 0 (before treatment), week 12 (after treatment) and week 36 (following up). Every time the participants receive the fMRI scan, they will be asked to finish the clinical scales. The primary outcome will be the change in the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) total score from baseline to week 12 and week 36. Secondary outcomes will include the changes of Hospital Anxiety and Depression Scale, International Prostate Symptom Score, International Index of Erectile Function, Self-Esteem Scale, Social Support Rating Scale and Numeric Rating Scale and brain functional activated or inactivated regions.

ELIGIBILITY:
Inclusion Criteria:

(1)The clinical diagnosis of CP/CPPS is exclusionary diagnosis.The main steps of diagnosing CP/CPPS are follwing: T

1. he chief complaint is long-term recurrent pain or discomfort of lumbosacral and perianal distension in the lower abdomen of the external perineum genital area and the superior pubic area (more than 3 months).
2. Bacterial prostatitis will be eliminated by routine culture of prostatic fluid and urine culture before and after prostatic massage.
3. Urinary tract infection will be ruled out by routine urinalysis and sediment examination.

(2)Total score of NIH-CPSI ≥ 15.

Exclusion Criteria:

The participants would be excluded if they got any acute or chronic infectious disease, other chronic pain diseases, internal organic diseases, history of malignant tumors, and chronic diseases that might contribute to peripheral nerve injury like diabetes mellitus and hypertension.

Prostate changes will be observed by prostate ultrasound and other urogenital and pelvic space-occupying lesions will be excluded.

Contraindications of fMRI scan like claustrophobia and denture implantation status are also considered.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To reduce the potential impact of senile brain atrophy, aged from 20 to 50 years volunteers were required.
Enrollment: 500 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-09-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in the NIH-CPSI total score at the end of week 12 and week 36 | week 0, week 12 and week 36
  The responder is defined as who has a decline of 6 or more than 6-point from baseline measured by using the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) , compared with the baseline in week 0.It is because a decline of at least 6 points in NIH-CPSI is acknowledged as the minimal clinically important difference. The NIH-CPSI is a self-assessment form with nine items, which the main components encompass pain with 4 items focused on location, severity and frequency, urinary function embracing one irritative item and one obstructive item, and quality of life impact with 3 items about the effect of symptoms on daily activities. The NIH-CPSI provides a systematized and unanimously accepted outcome measuring tool, and it is widely used in clinical trials, along with in the evidence-based evaluation of treatment effects.

SECONDARY OUTCOMES:
The alterations in brain of patients with CP/CPPS measured by fMRI when finishing the whole treatment | week 12
  By analysis of fMRI data, the potential alterations of treatment effect in brain will be concluded.
The alterations in brain of patients with CP/CPPS measured by fMRI in the following-up (24weeks after treatment) | week 36
  By analysis of fMRI data, the potential alterations of recurrence in brain will be concluded.
the change from baseline in NIH-CPSI subscales | week 0, week 12, week 36
  The alterations of NIH-CPSI subscales will provide the certain efficacy in the symptoms of CP/CPPS.
the change from baseline in the International Prostate Symptom Score (IPSS) | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of lower urinary tract symptoms.To detailly describe the symptoms of lower urinary tract, except for the NIH-CPSI, we will independently apply the International Prostate Symptom Score (IPSS). The IPSS covers seven symptom questions and one health-related quality of life (QoL) question.
the change from baseline in the Visual Analogue Scale (VAS) | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of pain.For pain assessment, the Numeric Rating Scale (NRS) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity and severity of pain.
the change from baseline in the Self-Esteem Scale (SES). | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of internal self esteem. In 1965, the Self-Esteem Scale (SES) was initially designed to assess adolescents' overall feelings of self-worth and self-acceptance by Rosenberg. The SES contains five positive and five negative items, which is a widely used and well validated measurement with good psychometric properties.
the change from baseline in the Social Support Rating Scale (SSRS) | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of external social support.The Social Support Rating Scale (SSRS) is a questionnaire with 10 items which consists of objective support (3 items), subjective support (4 items) and the utilization of social support (3 items), which assist to evaluate the characteristics of social support and its association with mental health level, mental illness and various physical diseases. The higher score, the more social support.
the change from baseline in the Quality of Life（QoL) | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of subjective life quality feeling. In patients with prostatic diseases, this score is mainly used to evaluate the impact of urination symptoms on quality of life, ranging from very good to very painful, with 0-6 points, to understand the subjective feelings of patients on the level of lower urinary tract symptoms, mainly concerned with the degree of distress caused by lower urinary tract symptoms and whether they can tolerate them. This score is always used within IPSS.
the change from baseline in NIH-CPSI | week 0, week 12, week 36
  These changes will reveal the efficacy of acupuncture in the aspect of symptoms of CP/CPPS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Acupuncture, LongHua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Chen J, Zhang H, Niu D, Li H, Wei K, Zhang L, Yin S, Liu L, Zhang X, Zhang M, Liang C. The risk factors related to the severity of pain in patients with Chronic Prostatitis/Chronic Pelvic Pain Syndrome. BMC Urol. 2020 Oct 7;20(1):154. doi: 10.1186/s12894-020-00729-9. PMID 33028277
- [Background] Krieger JN, Nyberg L Jr, Nickel JC. NIH consensus definition and classification of prostatitis. JAMA. 1999 Jul 21;282(3):236-7. doi: 10.1001/jama.282.3.236. No abstract available. PMID 10422990
- [Background] Zhong YM, Luo XC, Chen Y, Lai DL, Lu WT, Shang YN, Zhang LL, Zhou HY. Acupuncture versus sham acupuncture for simple obesity: a systematic review and meta-analysis. Postgrad Med J. 2020 Apr;96(1134):221-227. doi: 10.1136/postgradmedj-2019-137221. Epub 2020 Feb 3. PMID 32015189
- [Background] Hopton A, MacPherson H. Acupuncture for chronic pain: is acupuncture more than an effective placebo? A systematic review of pooled data from meta-analyses. Pain Pract. 2010 Mar-Apr;10(2):94-102. doi: 10.1111/j.1533-2500.2009.00337.x. Epub 2010 Jan 8. PMID 20070551
- [Background] Passavanti MB, Pota V, Sansone P, Aurilio C, De Nardis L, Pace MC. Chronic Pelvic Pain: Assessment, Evaluation, and Objectivation. Pain Res Treat. 2017;2017:9472925. doi: 10.1155/2017/9472925. Epub 2017 Nov 20. PMID 29359045
- [Background] Bhatt RR, Gupta A, Mayer EA, Zeltzer LK. Chronic pain in children: structural and resting-state functional brain imaging within a developmental perspective. Pediatr Res. 2020 Dec;88(6):840-849. doi: 10.1038/s41390-019-0689-9. Epub 2019 Dec 2. PMID 31791045
- [Background] Ge S, Hu Q, Guo Y, Xu K, Xia G, Sun C. Potential Alterations of Functional Connectivity Analysis in the Patients with Chronic Prostatitis/Chronic Pelvic Pain Syndrome. Neural Plast. 2021 May 7;2021:6690414. doi: 10.1155/2021/6690414. eCollection 2021. PMID 34035803
- [Background] Park JJ. Developing and validating a sham acupuncture needle. Acupunct Med. 2009 Sep;27(3):93. doi: 10.1136/aim.2009.001495. No abstract available. PMID 19734377